CLINICAL TRIAL: NCT02615288
Title: Impact of High Dose Vitamin D3 Supplementation in Treatment of Crohn's Disease in Remission: A Randomized Double-blind Controlled Study
Brief Title: High Dose Vitamin D3 in Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Association of Gastroenterology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-038
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Crohn's Disease
Keywords: Vitamin D
MeSH Terms: conditions — Crohn Disease | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose Vitamin D3 (10,000 IU daily) (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3
- Low Dose Vitamin D3 (1000 IU daily) (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3

SUMMARY:
This is a randomized, double-blind placebo-controlled trial of high dose vitamin D3 at 10,000 International Units (IU) daily compared to low dose at 1000 IU daily in patients with Crohn's disease in remission.

DETAILED DESCRIPTION:
In patients with Crohn's disease in remission, the investigators hypothesized higher doses of vitamin D would more effectively improve 25-hydroxy(OH)-vitamin D levels and would be tolerated well without side effects of hypercalcemia. The investigators also wanted to explore whether higher doses could reduce the clinical relapse rate of patients with Crohn's disease in remission, and if higher doses of vitamin D3 could improve depression and anxiety symptoms. In order to determine if there is benefit from high-dose vitamin D3, the investigators designed a pilot randomized double-blind controlled trial comparing doses of oral vitamin D3 at 10,000 IU daily to 1000 IU daily.

ELIGIBILITY:
Inclusion Criteria:

* a prior diagnosis of Crohn's disease in clinical remission for at least 28 days with a Harvey-Bradshaw index less than or equal to 4
* All maintenance therapies for Crohn's disease will be required to be at stable dose for at least 3 months before randomization, with no systemic steroid therapy within 4 weeks.
* Vitamin D supplements will be discontinued at least 6 weeks before randomization.

Exclusion Criteria:

* Women of child bearing potential who are considering pregnancy during the study period, currently pregnant, or unwilling to use contraception to avoid pregnancy
* Participants with renal insufficiency (serum creatinine greater than 150 umol/L), sarcoidosis, hyperparathyroidism, malignancy, or any other disorder that may lead to hypercalcemia
* Patients with short-gut syndrome or a serum albumin less than 32 g/L
* Concomitant therapy with thiazide diuretics, barbiturates, digitalis, or supplemental products containing vitamin D

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Improvement in 25-OH vitamin D level | One year

SECONDARY OUTCOMES:
Clinical Remission (defined as Harvey-Bradshaw index <=4) | One year
  Number of patients who maintain clinical remission
Improvement in Depression scores (measured by Hospital Anxiety and Depression Scale (HADS)) | One year
  Number of patients who achieve significant improvement in HADS (reduction of 2 or more)
Improvement in C-reactive protein | One year
  Comparison of C-reactive protein levels in high and low dose vitamin D3 groups
Adverse events | One year
  Number of patients with treatment-related adverse events, including death, hypercalcemia, and hospitalization, as well as minor adverse events

REFERENCES:
- [Derived] Narula N, Cooray M, Anglin R, Muqtadir Z, Narula A, Marshall JK. Impact of High-Dose Vitamin D3 Supplementation in Patients with Crohn's Disease in Remission: A Pilot Randomized Double-Blind Controlled Study. Dig Dis Sci. 2017 Feb;62(2):448-455. doi: 10.1007/s10620-016-4396-7. Epub 2016 Dec 14. PMID 27975236